CLINICAL TRIAL: NCT03430245
Title: Pilot Study to Evaluate VelaShape III & UltraShape Power Combined Treatment for Thigh Circumference Reduction
Brief Title: VelaShape III & UltraShape Power for Thigh Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF24451
Record Dates: First submitted 2018-01-24; First posted 2018-02-12 (Actual); Results first posted 2019-12-26 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Circumference Reduction
Keywords: Circumference reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VelaShape III & UltraShape Power (Experimental): VelaShape III treatment with radiofrequency, infrared and massage combined with UltraShape Power treatment, using pulsed, focused ultrasound treatment.
  Interventions: Device: VelaShape III; Device: UltraShape Power

INTERVENTIONS:
Device: VelaShape III — The VelaShape III device combines controlled infrared (IR) light and conducted bipolar radiofrequency (RF) energies with vacuum.
Device: UltraShape Power — The UltraShape Power device uses focused ultrasound energy for lipolysis (breakdown of fat) via a non-thermal mechanism of action.

SUMMARY:
Prospective, one-arm, baseline-controlled pilot study for the evaluation of the VelaShape III combined with UltraShape Power treatment for non-invasive circumference reduction to the thighs.

DETAILED DESCRIPTION:
Eligible subjects will receive 3 bi-weekly treatments to the thighs at 2-week intervals, with the VelaShape III and UltraShape Power devices according to the study protocol.

Each subject will return for 3 follow up visits: four weeks (4wk FU), 8 weeks (8wk FU) and 12 weeks (12wk FU) after the last treatment (Tx.3), for total expected study duration of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Female and male subjects, 18 and 60 years of age at the time of enrollment.
3. Fitzpatrick Skin Type I to VI.
4. Fat thickness of at least 1.5 cm (measured by calibrated caliper).
5. BMI interval: 22 ≤ BMI ≤ 30 (normal to overweight, but not obese).
6. Female subjects must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
7. In addition, negative urine pregnancy test as tested before each treatment and at the last visit for women with child-bearing potential (e.g. not menopausal).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations.

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism.
2. Known hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease.
3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone.
6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction.
7. Previous body contouring procedures in the treatment area within 12 months.
8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing.
9. Known photosensitivity.
10. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
11. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area.
12. Very poor skin quality (i.e., severe laxity).
13. Abdominal wall diastasis or hernia on physical examination.
14. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months.
15. Obesity (BMI > 30).
16. Pregnant, childbirth within the last 12 months or breastfeeding women.
17. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study.
18. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months).
19. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration).
20. Abdominal fat thickness lower than 2.5 cm after strapping.
21. Participation in another clinical study within the last 6 months.
22. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Laser & Surgery Specialist of NY/NJ, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coleman WP 3rd, Coleman W 4th, Weiss RA, Kenkel JM, Ad-El DD, Amir R. A Multicenter Controlled Study to Evaluate Multiple Treatments With Nonthermal Focused Ultrasound for Noninvasive Fat Reduction. Dermatol Surg. 2017 Jan;43(1):50-57. doi: 10.1097/DSS.0000000000000918. PMID 28009680

RESULTS

PARTICIPANT FLOW:
Groups:
- VelaShape III & UltraShape Power: Subjects received 3 biweekly treatments to the thighs with the VelaShape III and UltraShape Power devices.
  The VelaShape III device combines controlled infrared (IR) light and conducted bipolar radiofrequency (RF) energies with vacuum.
  The UltraShape Power device uses focused ultrasound energy for lipolysis (breakdown of fat) via a non-thermal mechanism of action.
Period: Overall Study
Arm/Group | VelaShape III & UltraShape Power
Started | 16
Completed | 9 (6 subjects withdrew from study due to lengthy treatment. Treatment protocol amended.)
Not Completed | 7
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Subjects treated with VelaShape III and UltraShape Power
Units Other Than Participants: Number of thighs
Arm/Group | VelaShape III & UltraShape Power
Number analyzed (Participants) | 16
Number analyzed (Number of thighs) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Mean thigh circumference [Mean (Standard Deviation); unit: centimeter] — Collected using a measuring tape at thigh midline
  centimeter | 62.1 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Circumference Change in the Thighs at the 12-week Follow-up Compared to Baseline Measurements
Description: Circumference change of thigh midline post combined VelaShape III and UltraShape Power treatments. Negative change represent reduction in thigh circumference.
Time Frame: At 12 weeks after the third treatment (week 16) for each subject
Population: 6 subjects were initially treated, but then were lost to follow-up during the period when the treatment protocol was amended. One other subject was lost to follow-up after three treatments because she was unable to come in for visits due to work schedule
Measure: Mean (Standard Deviation); unit: centimeter
Units Other Than Participants: Number of thighs
Groups:
- VelaShape III & UltraShape Power: Subjects left and right thighs were each treated with both VelaShape III and UltraShape Power, a combined treatment.
Arm/Group | VelaShape III & UltraShape Power
Number analyzed (Participants) | 9
Number analyzed (Number of thighs) | 18
centimeter | -2.8 (1.8)

2. Secondary Outcome: Change in the Thighs Circumference at Each Treatment Visit Post Baseline and at The 4 and 8 Week Follow-up Visits
Description: The thighs circumference change (at midline) after combined treatment with VelaShape III and UltraShape Power treatments compared to baseline.
  The changed of thighs circumference was calculated at 2, 4, 8 and 12 weeks after baseline (which are second treatment , third treatment, 4 and 8 week follow-up visits, respectively).
  Negative change represent reduction in thigh circumference.
Time Frame: At 2, 4, 8 and 12 weeks after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeter
Units Other Than Participants: Number of Thighs
Arm/Group | VelaShape III & UltraShape Power
Number analyzed (Participants) | 10
Number analyzed (Number of Thighs) | 20
centimeter
  Circumference change at the second treatment | -0.4 (0.6)
  Circumference change at the third treatment | -0.8 (0.7)
  Circumference change at 8 weeks after baseline: number analyzed (Participants) | 9
  Circumference change at 8 weeks after baseline: number analyzed (Number of Thighs) | 18
  Circumference change at 8 weeks after baseline | -1.8 (0.8)
  Circumference change at 12 weeks after baseline: number analyzed (Participants) | 9
  Circumference change at 12 weeks after baseline: number analyzed (Number of Thighs) | 18
  Circumference change at 12 weeks after baseline | -2.2 (1.6)

3. Secondary Outcome: Investigator Satisfaction
Description: Investigator satisfaction assessment performed independently, using a 5- point Likert scale questionnaire from 2=very satisfied to -2=very unsatisfied at each follow-up visits (4, 8 and 12 weeks after the last treatment)
Time Frame: At 4, 8 and 12 weeks follow-up visits
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | VelaShape III & UltraShape Power
Number analyzed (Participants) | 9
Participants
  Investigator satisfaction at 4 week follow-up: (-2) Very unsatisfied | 0
  Investigator satisfaction at 4 week follow-up: (-1) Unsatisfied | 0
  Investigator satisfaction at 4 week follow-up: (0) No Opinion | 0
  Investigator satisfaction at 4 week follow-up: (1) Satisfied | 5
  Investigator satisfaction at 4 week follow-up: (2) Very satisfied | 4
  Investigator satisfaction at 8 week follow-up: (-2) Very unsatisfied | 0
  Investigator satisfaction at 8 week follow-up: (-1) Unsatisfied | 0
  Investigator satisfaction at 8 week follow-up: (0) No Opinion | 0
  Investigator satisfaction at 8 week follow-up: (1) Satisfied | 4
  Investigator satisfaction at 8 week follow-up: (2) Very satisfied | 5
  Investigator satisfaction at 12 week follow-up: (-2) Very unsatisfied | 0
  Investigator satisfaction at 12 week follow-up: (-1) Unsatisfied | 0
  Investigator satisfaction at 12 week follow-up: (0) No Opinion | 0
  Investigator satisfaction at 12 week follow-up: (1) Satisfied | 2
  Investigator satisfaction at 12 week follow-up: (2) Very satisfied | 7

4. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction assessment performed independently, using a 5- point Likert scale questionnaire from 2=very satisfied to -2=very unsatisfied at each follow-up visits (at 4, 8 and 12 weeks after the last treatment visit).
Time Frame: At 4, 8 and 12 week follow-up visits
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | VelaShape III & UltraShape Power
Number analyzed (Participants) | 9
Participants
  Subject satisfaction at 4 week follow-up: (-2) Very unsatisfied | 0
  Subject satisfaction at 4 week follow-up: (-1) Unsatisfied | 0
  Subject satisfaction at 4 week follow-up: (0) No Opinion | 0
  Subject satisfaction at 4 week follow-up: (1) Satisfied | 3
  Subject satisfaction at 4 week follow-up: (2) Very satisfied | 6
  Subject satisfaction at 8 week follow-up: (-2) Very unsatisfied | 0
  Subject satisfaction at 8 week follow-up: (-1) Unsatisfied | 0
  Subject satisfaction at 8 week follow-up: (0) No Opinion | 1
  Subject satisfaction at 8 week follow-up: (1) Satisfied | 3
  Subject satisfaction at 8 week follow-up: (2) Very satisfied | 5
  Subject satisfaction at 12 week follow-up: (-2) Very unsatisfied | 0
  Subject satisfaction at 12 week follow-up: (-1) Unsatisfied | 0
  Subject satisfaction at 12 week follow-up: (0) No Opinion | 0
  Subject satisfaction at 12 week follow-up: (1) Satisfied | 2
  Subject satisfaction at 12 week follow-up: (2) Very satisfied | 7

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected is from treatment visit until 12 weeks follow-up (16 weeks post baseline) treatment
Description: The number and severity of adverse events following each treatment, with combined Velashape III and Ultrashape Power for the thighs, were evaluated at each of the three biweekly visits and at the 4, 8 and 12 weeks following the treatment.
Arm/Group | VelaShape III & UltraShape Power
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VelaShape III & UltraShape Power (N=16)
Blistering (Skin and subcutaneous tissue disorders) | 1 (1) — Patient developed 2 blisters on left thigh at the day after the second treatment. Subject advised to keep area clean & covered and to temporarily discontinue treatments. The blisters recovered without intervention.

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03430245/Prot_SAP_000.pdf